CLINICAL TRIAL: NCT07018908
Title: Effect of Intake of Dehydrated Nopal Powder From Highly Mature Cladodes (Opuntia Ficus-indica) on the Lipid Profile of Overweight or Obese Adults. A Randomized Controlled Trial.
Brief Title: Effect of Intake of Dehydrated Nopal Powder From Highly Mature Cladodes on the Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Querétaro (Other)
Responsible Party: Principal Investigator, Maria de los Angeles Aguilera Barreiro, Director and Principal Investigator, Universidad Autónoma de Querétaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCN-10310
Record Dates: First submitted 2025-05-25; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Obesity; Dyslipidemia
Keywords: Opuntia ficus-indica; dyslipidemia; overweight; obesity; diet
MeSH Terms: conditions — Overweight; Obesity; Dyslipidemias | interventions — Dietary Supplements; Control Groups

STUDY DESIGN:
Intervention Model Description: Group I (first arm): 5 g of dehydrated nopal + normocaloric diet. Group II (second arm): 15 g of dehydrated nopal + normocaloric diet. Group III (third arm): normocaloric diet only (control or comparison group).
  This design allows for the comparison of the effects of different doses or treatments (in this case, different amounts of nopal) against a control (the diet alone).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (first arm): 5 g of dehydrated nopal + normocaloric diet. (Active Comparator): Supplementation: 5 g of dehydrated nopal (2.47 g of fiber per day), reconstituted in water, taken before breakfast. Diet: 27.53 g of fiber per day, Normocaloric diet: Carbohydrates: 55%, Lipids 25% and Proteins 20%
  Interventions: Dietary Supplement: supplementation with 5 g dehydrated nopal powder from highly mature cladodes
- Group II (second arm): 15 g of dehydrated nopal + normocaloric diet. (Active Comparator): Supplementation: 15 g of dehydrated nopal (7.42 g of fiber per day), reconstituted in water, taken before breakfast and at night. Diet: 22.58 g of fiber per day, Normocaloric diet: Carbohydrates 55%, Lipids 25% and Proteins 20%
  Interventions: Dietary Supplement: supplementation with 15 g dehydrated nopal powder from highly mature cladodes
- Group III (third arm): normocaloric diet only (control or comparison group). (Other): No dehydrated nopal or placebo. 30 g of fiber per day Normocaloric diet Carbohydrates 55%, Lipids 25% and Proteins 20%
  Interventions: Other: Control Group (only diet)

INTERVENTIONS:
Dietary Supplement: supplementation with 5 g dehydrated nopal powder from highly mature cladodes — Group I received 5 g of dehydrated Opuntia ficus-indica cladodes plus the standard normocaloric diet for dyslipidemia.
  Arms: Group I (first arm): 5 g of dehydrated nopal + normocaloric diet.
Dietary Supplement: supplementation with 15 g dehydrated nopal powder from highly mature cladodes — Group II received 15 g plus the diet, and Group III followed only the diet.
  Arms: Group II (second arm): 15 g of dehydrated nopal + normocaloric diet.
Other: Control Group (only diet) — No dehydrated nopal or placebo. Diet: 30 g of fiber per day Normocaloric diet Carbohydrates 55%, Lipids 25% and Proteins 20%
  Arms: Group III (third arm): normocaloric diet only (control or comparison group).

SUMMARY:
Background: Opuntia ficus-indica is a plant from the cactus family (Cactaceae) that is widespread and of great economic importance in Mexico. It has been consumed as food since pre-Hispanic times and is currently considered a nutraceutical. In this study, the effect of consumption of dehydrated nopal powder from highly mature cladodes (Opuntia ficus-indica) on the lipid profile of overweight or obese patients diagnosed with dyslipidemia was investigated. Methods: A 3-month prospective clinical trial was conducted in 35 overweight or obese patients with dyslipidemia. The sample was divided into three groups with a daily intake of 30 g of dietary fiber: Group I received 5 g of dehydrated Opuntia ficus-indica cladodes plus the standard normocaloric diet for dyslipidemia, Group II received 15 g plus the diet, and Group III followed only the diet.

ELIGIBILITY:
Inclusion Criteria:

* Participants with dyslipidemia, confirmed by lipid meas-urement in blood chemistry
* overweight or obesity
* A cardiovascular risk factor associated with abdominal obesity

Exclusion Criteria:

* Patients with a suspected diagnosis of primary dyslipidemia
* Diabetes
* Hypertension
* Thyroid disease were excluded from the study
* Patients with complex or severe disease such as heart failure, liver or kidney disease
* Pregnant or lactating women
* Indidividuals taking lipid-modifying drugs or hormone replacement therapy - Patients with gastrointestinal problems and deficiencies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Blood lipid levels | From enrollment to the end of treatment at 12 weeks
  A blood sample (3 ml) was taken from the patients after fasting for 12 hours, then prepared for subsequent analysis by an enzymatic method. The Clinical 50 VWR cen-trifuge ® was used for sample preparation and the Roche Cobas C 111 ® kit for lipid analysis of the samples. These analyses were performed in duplicate. Comparison of supplementation with dehydrated nopal powder from highly mature cladodes, by group, in initial and final values of the lipid profile: Total cholesterol; LDL, Low-density lipoproteins; HDL, High-density lipoproteins; TGL, Tri-glycerides.

CONTACTS AND LOCATIONS:
Locations (1):
- Autonomous University of Queretaro, Juriquilla, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: No